CLINICAL TRIAL: NCT04279184
Title: Urinary Incontinence and Endocrine Factors.
Brief Title: Urinary Incontinence and Endocrine Factors. A Part of Lolland-Falster Health Study (LOFUS).
Acronym: EFUI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nykøbing Falster County Hospital (Other)
Collaborators: Region Zealand (Other); Zealand University Hospital (Other); University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: SJ-493
Record Dates: First submitted 2020-01-16; First posted 2020-02-21 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Urinary Incontinence; Diabetes; Thyroid Diseases
MeSH Terms: conditions — Urinary Incontinence; Diabetes Mellitus; Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Previous studies have shown an increase in the prevalence of urgency and urgency incontinence in women with diabetes. Regarding the condition urinary stress incontinence, the literature is diverted.

The purpose of the PhD project is investigate the prevalence of urinary incontinence and the association to diabetes and thyroid disease in a mainly rual population in Lolland and Falster. Further to investigate if there is any difference in the bladder function in incontinent women with and without diabetes.

Psychometric validation of the questionnaire used to assess urinary incontinence was also performed.

ELIGIBILITY:
Inclusion Criteria:

* woman
* 18 years or above
* participating i The Lolland-Falster Health Study (NCT02482896)

Exclusion Criteria:

* male
* below 18 years
* non-participating i The Lolland-Falster Health Study

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The population of Lolland and Guldborgsund municipalities in Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence of urinary incontinence | 4 years
  Assess by self-administered questionnaire and register data. Cross-sectional, measure once. The questionnaire International Consultation on Incontinence Questionnaire - Urinary Incontinence Short form (ICIQ-UI SF) was used to assess urinary incontinence (UI). It consist of six questions, and the score of three of the questions (assessing frequency of UI, volume of leak and bother) sums up to a total score. It ranges between 0-21 where 0 is no incontinence and a higher score indicates more severe symptoms of UI. The inclusion of participants are over a period of four years.
Psychometric validation of ICIQ-UI SF (questionnaire used to assess urinary incontinence) | 2 years
  We investigated the predictive validity, internal consistency, patient-interview agreement, construct validity, test-retest reliability, and sensitivity to change for the ICIQ-UI SF.

SECONDARY OUTCOMES:
Association between urinary incontinence and diabetes | 4 years
  Assess by self-administered questionnaire and register data. Cross-sectional, measure once. The inclusion of participants are over a period of four years.
Participants demographics | 4 years
  Assess by self-administered questionnaire and register data. Cross-sectional, measure once. The inclusion of participants are over a period of four years.
Objective characterization of urinary incontinence in women with and without diabetes | 2 years
  Assess by urodynamics studies. Description of type of urinary incontinence, first sensation (ml), normal desire (ml), urgency (ml), max capacity (ml) and PVR (ml). Measured once for each participants. Data collected over a period of two years.

CONTACTS AND LOCATIONS:
Overall Officials: Helga Gimbel, Principal Investigator — Zealand University Hospital
Locations (1):
- Randi Jepsen, Nykøbing Falster, Danmark, Denmark